CLINICAL TRIAL: NCT00346970
Title: Randomized Clinical Trial to Study the Effect of Extended Release Niacin on Endothelial Function, Oxidative Stress and Endothelial Progenitor Cells in Patients With the Metabolic Syndrome.
Brief Title: The High Density Lipoprotein and Endothelial Function, Niacin and Nitric Oxide Study (The High-Ennd Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-005694-30
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; High Density Lipoprotein; Extended-Release Niacin; Endothelial Function; Endothelial Progenitor Cells
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): Extended-release Niacin
  Interventions: Drug: Extended-Release Niacin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Extended-Release Niacin — Extended-Release Niacin tablets week 1-4 500 mg/d week 4-8 1000 mg/d week 9-12 1500 mg/d
  Arms: 1
Drug: Placebo — Placebo tablets
  Arms: 2

SUMMARY:
The aim of the present study is to characterize novel mechanisms whereby HDL may exert potent vasculoprotective effects independent of reverse cholesterol transport, in particular the effect of HDL on the regulation of the vascular NAD(P)H oxidase enzyme system, a major vascular source of superoxide, known to be important for endothelial dysfunction. In addition, the present study will characterize the effect of HDL on endothelial progenitor cell (EPC) mobilization, nitric oxide production and in vivo regenerative capacity.

ELIGIBILITY:
Inclusion Criteria:

* Statin treatment for at least 3 weeks
* Reduced HDL: < 40 mg/dL (1.03 mmol/L) in men or < 50 mg/dL (1.29 mmol/L) in women
* Plus TWO of the following (thereby defining the patients to have metabolic syndrome (Grundy et al.; Circulation 2005)):
* Elevated waist circumference: ≥ 102 cm (≥ 40 inches) in men or ≥ 88 cm (≥ 35 inches) in women
* Elevated triglycerides: ≥ 150 mg/dL (1.7 mmol/L
* Elevated blood pressure: ≥ 130 mmHg systolic blood pressure or ≥ 80 mmHg diastolic blood pressure or anti-hypertensive treatment
* Elevated fasting glucose: ≥ 100 mg/dL or on drug treatment for elevated fasting glucose

Exclusion Criteria:

* Hypersensitivity to niacin
* Active liver disease or impaired liver function
* Persistent elevation of transaminases
* Cholestasis
* Gastric ulcer
* Acute coronary syndrome
* Gout
* Pregnancy, lactation
* Active infections
* Cancer
* Untreated concomitant diseases
* Renal insufficiency or renal failure
* Hypothyreosis
* Alcoholism
* Myopathies
* Muscle pain under therapy with fibrates or statins
* Hereditary muscle diseases in family history

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Antioxidative Properties of Endothelial Progenitor Cells | 3 months
FDD | 3 months

SECONDARY OUTCOMES:
High Density Lipoprotein (HDL) Elevation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Drexler, MD, Study Director — Hannover Medical School; Ulf Landmesser, MD, Principal Investigator — Hannover Medical School; Sajoscha A Sorrentino, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Sorrentino SA, Besler C, Rohrer L, Meyer M, Heinrich K, Bahlmann FH, Mueller M, Horvath T, Doerries C, Heinemann M, Flemmer S, Markowski A, Manes C, Bahr MJ, Haller H, von Eckardstein A, Drexler H, Landmesser U. Endothelial-vasoprotective effects of high-density lipoprotein are impaired in patients with type 2 diabetes mellitus but are improved after extended-release niacin therapy. Circulation. 2010 Jan 5;121(1):110-22. doi: 10.1161/CIRCULATIONAHA.108.836346. Epub 2009 Dec 21. PMID 20026785